CLINICAL TRIAL: NCT00252512
Title: Effectiveness of Contingency Management in VA Addictions Treatment
Brief Title: The Effect of a Contingency Management Intervention on Substance Use
Acronym: REAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 03-120
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2014-08-29 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Substance Use Disorders
Keywords: Contingency management interventions; Substance use disorders treatment; Treatment effectiveness; Randomized clinical trial; Behavioral research
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contingency Management (Experimental): Participants complete urine and breath screens 2 times per week for 8 weeks. If urine and breath screens are negative, they receive a chance to draw tokens from a bowl. Some tokens are social reinforcement. Others have monetary value.
  Interventions: Behavioral: Contingency Management
- Placebo (Placebo Comparator): Participants complete urine and breath screens 2 times per week for 8 weeks with no reinforcement for negative results.
  Interventions: Other: Placebo

INTERVENTIONS:
Behavioral: Contingency Management — Participants complete urine and breath screens 2 times per week for 8 weeks. If urine and breath screens are both negative, the participant receives a chance to draw tokens from a bowl. Some tokens are social reinforcement (Good Job!). Other have monetary value.
  Arms: Contingency Management
Other: Placebo — Participants complete urine and breath screens 2 times per week for 8 weeks with no reinforcement for negative results.
  Arms: Placebo

SUMMARY:
Contingency management interventions involve providing a tangible reward for progress toward treatment goals. The purpose of this study is to determine whether a contingency management intervention added to usual care leads to improved attendance and decreased substance use in patients attending outpatient substance use disorders treatment.

DETAILED DESCRIPTION:
Design: This will be a randomized, controlled trial. 360 veterans presenting for specialty substance use disorders treatment at the Minneapolis VAMC and the VA Puget Sound Health Care System will be randomly assigned to 8 weeks of Usual Care or Usual Care plus Contingency Management. Minimal exclusion criteria include primary cannabis dependence, primary opioid dependence, screening positive for pathological gambling, serious psychiatric symptoms or suicide risk. Randomization will be stratified by site and primary substance use disorder (alcohol or stimulant). All participants will meet with a research assistant twice per week to submit urine drug and breath alcohol samples. Participants randomized to the contingency management interventions will have the opportunity to draw tokens (with replacement) from a bowl each time they submit negative urine drug and breath alcohol screens. The number of drawings allowed escalates with continuous weeks of negative screens or returns to baseline if screens are positive or missed. Half of the 500 tokens will result in social reinforcement ("Good Job!"). The remainder will earn a VA canteen voucher worth monetary value. Follow-up assessments occur 2, 6, and 12 months after enrollment into the study. Primary outcomes measures include number of days with negative urine drug and breath alcohol screens during the intervention phase, days of treatment attendance during the intervention phase, and percent days abstinent on the Timeline Follow-Back interview at follow-up assessments. Secondary outcomes include a brief assessment of employment, housing, legal, and psychiatric status, and administrative data on VA service utilization. A process evaluation and an economic analysis are included.

ELIGIBILITY:
Inclusion Criteria:

* veterans presenting for outpatient substance use disorders treatment with a diagnosis of alcohol, cocaine, amphetamine, or methamphetamine dependence

Exclusion Criteria:

* primary cannabis dependence
* primary opioid dependence
* severe psychiatric symptoms
* suicide risk
* positive history or screen for pathological gambling
* lacking transportation or living too far away to attend twice per week research appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2007-05; Primary Completion 2010-01 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hildi J. Hagedorn, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (2):
- United States (2):
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

REFERENCES:
- [Result] Hagedorn HJ, Noorbaloochi S, Simon AB, Bangerter A, Stitzer ML, Stetler CB, Kivlahan D. Rewarding early abstinence in Veterans Health Administration addiction clinics. J Subst Abuse Treat. 2013 Jul;45(1):109-17. doi: 10.1016/j.jsat.2013.01.006. Epub 2013 Feb 28. PMID 23453480
- [Result] Hagedorn HJ, Stetler CB, Bangerter A, Noorbaloochi S, Stitzer ML, Kivlahan D. An implementation-focused process evaluation of an incentive intervention effectiveness trial in substance use disorders clinics at two Veterans Health Administration medical centers. Addict Sci Clin Pract. 2014 Jul 9;9(1):12. doi: 10.1186/1940-0640-9-12. PMID 25008457
- [Result] Hagedorn HJ, Noorbaloochi S, Bangerter A, Stitzer ML, Kivlahan D. Health care cost trajectories in the year prior to and following intake into Veterans Health Administration outpatient substance use disorders treatment. J Subst Abuse Treat. 2017 Aug;79:46-52. doi: 10.1016/j.jsat.2017.05.013. Epub 2017 May 25. PMID 28673526

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants withdrew from participation after random assignment to the placebo condition and did not start the intervention.
Period: Intervention
Arm/Group | Contingency Management | Placebo
Started | 165 | 165
Completed | 136 | 134
Not Completed | 29 | 31
Period: Six Month Follow up
Arm/Group | Contingency Management | Placebo
Started | 136 | 134
Completed | 132 | 122
Not Completed | 4 | 12
Period: 12 Month Follow up
Arm/Group | Contingency Management | Placebo
Started | 132 | 122
Completed | 123 | 121
Not Completed | 9 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Contingency Management | Placebo | Total
Number analyzed (Participants) | 165 | 165 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (9.7) | 49.5 (8.1) | 49.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 160 | 163 | 323
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 162 | 158 | 320
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 60 | 53 | 113
  White | 90 | 98 | 188
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 14 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 165 | 165 | 330

OUTCOME MEASURES:

1. Primary Outcome: Number of Negative Breath Alcohol and Urine Drug Screens Out of Possible 16
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: negative alcohol and drug screens
Arm/Group | Contingency Management | Placebo
Number analyzed (Participants) | 165 | 165
negative alcohol and drug screens | 11.93 (4.67) | 10.39 (5.18)
Statistical Analysis 1: Comparison: Contingency Management vs Placebo; Test type: Superiority; p < .001, GEE full factorial modeling — Above is calculated p value, a priori threshold for significance set at <.05

2. Secondary Outcome: Psychiatric Status
Description: Kessler Psychological Distress Scale (K10) - score range 10 to 50.
  * score under 20 are likely to be well
  * score 20-24 are likely to have mild psychological distress
  * score 25-29 are likely to have moderate psychological distress
  * score 30 and over are likely to have a severe psychological distress
Time Frame: 8 weeks, 6 months, 12 months
Population: Fewer participants completed 6 and 12 month follow-up assessments than completed 8 week assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Contingency Management | Placebo
Number analyzed (Participants) | 134 | 133
units on a scale
  8 week outcomes | 20.87 (6.42) | 18.90 (6.68)
  6 month outcomes: number analyzed (Participants) | 131 | 120
  6 month outcomes | 20.64 (8.31) | 20.19 (7.42)
  12 month outcomes: number analyzed (Participants) | 121 | 121
  12 month outcomes | 21.06 (8.23) | 19.07 (7.46)
Statistical Analysis 1: Comparison: Contingency Management vs Placebo; 8 week analysis; Test type: Superiority; p = .015, t-test, 2 sided — a priori threshold of <.05
Statistical Analysis 2: Comparison: Contingency Management vs Placebo; 6 month analysis; Test type: Superiority; p = 0.45, t-test, 2 sided — a priori threshold of <.05
Statistical Analysis 3: Comparison: Contingency Management vs Placebo; 12 month analysis; Test type: Superiority; p = .0497, t-test, 2 sided — a prior threshold of .05

3. Secondary Outcome: VHA Healthcare Service Utilization
Description: Cost of total healthcare utilization for six month period between baseline and 6 month follow up and six month period between 6 month and 12 month follow up.
Time Frame: Baseline to 6 month follow up and 6 month follow up to 12 month follow up.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Contingency Management | Placebo
Number analyzed (Participants) | 165 | 165
Dollars
  Total VHA healthcare costs: baseline-6 month f/up | 12744.44 (16321.11) | 16456.32 (28113.13)
  Total VHA healthcare costs: 6 month-12 month f/up | 8934.52 (13467.21) | 8386.94 (13667.40)
Statistical Analysis 1: Comparison: Contingency Management vs Placebo; Costs for period between 6 month follow-up and 12 month follow up; Test type: Superiority; p > .05, Estimation Equation mean modeling — a priori threshold <.05
Statistical Analysis 2: Comparison: Contingency Management vs Placebo; Costs for period between 6 month follow up and 12 month follow up; Test type: Superiority; p > .05, Estimating Equation mean modeling

4. Secondary Outcome: Housing
Description: Number of participants reporting stable housing (owned or rented house, apartment or room)
Time Frame: 8 week, 6 month and 12 month follow-ups
Population: Fewer participants completed 6 and 12 month follow-up assessments than completed 8 week follow up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Contingency Management | Placebo
Number analyzed (Participants) | 136 | 132
Participants
  Housing status at 8 weeks | 77 | 66
  Housing status at 6 months: number analyzed (Participants) | 132 | 121
  Housing status at 6 months | 80 | 91
  Housing at 12 months: number analyzed (Participants) | 123 | 120
  Housing at 12 months | 88 | 88
Statistical Analysis 1: Comparison: Contingency Management vs Placebo; Analysis for 8 week follow up; Test type: Superiority; p = .28, Chi-squared — a priori threshold <.05
Statistical Analysis 2: Comparison: Contingency Management vs Placebo; Analysis for 6 month follow up; Test type: Superiority; p = .013, Chi-squared — A priori threshold <.05
Statistical Analysis 3: Comparison: Contingency Management vs Placebo; Analysis for 12 month follow up; Test type: Superiority; p = .76, Chi-squared — A priori threshold <.05

5. Secondary Outcome: Legal Status
Description: Number of participants reporting detention or incarceration in the previous 30 days
Time Frame: 8 weeks, 6 month and 12 month follow ups
Population: Lower numbers of participants returned for 6 and 12 month follow up assessments compared to 8 week follow up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Contingency Management | Placebo
Number analyzed (Participants) | 136 | 134
Participants
  Legal status at 8 week follow-up | 3 | 2
  Legal status at 6 month follow-up: number analyzed (Participants) | 132 | 122
  Legal status at 6 month follow-up | 6 | 3
  Legal status at 12 month follow up: number analyzed (Participants) | 123 | 121
  Legal status at 12 month follow up | 3 | 7
Statistical Analysis 1: Comparison: Contingency Management vs Placebo; Analysis for 8 week follow-up; Test type: Superiority; p = .66, Chi-squared — A priori threshold <.05
Statistical Analysis 2: Comparison: Contingency Management vs Placebo; Analysis for 6 month follow up; Test type: Superiority; p = .37, Chi-squared — A priori threshold <.05
Statistical Analysis 3: Comparison: Contingency Management vs Placebo; Analysis for 12 month follow up; Test type: Superiority; p = .19, Chi-squared — a priori threshold <.05

6. Secondary Outcome: Employment Status
Description: Number of participants identifying themselves as unemployed.
Time Frame: 8 week, 6 month and 12 month follow up
Population: Fewer participants completed 6 and 12 month follow up assessments compared to 8 week follow up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Contingency Management | Placebo
Number analyzed (Participants) | 136 | 134
Participants
  Employment status at 8 week follow-up | 74 | 57
  Employment status at 6 month follow-up: number analyzed (Participants) | 132 | 122
  Employment status at 6 month follow-up | 51 | 49
  Employment status at 12 week follow-up: number analyzed (Participants) | 122 | 121
  Employment status at 12 week follow-up | 32 | 43
Statistical Analysis 1: Comparison: Contingency Management vs Placebo; Analysis for 8 week follow-up; Test type: Superiority; p = .05, Chi-squared — A priori threshold of <.05
Statistical Analysis 2: Comparison: Contingency Management vs Placebo; Analysis for 6 month follow-up; Test type: Superiority; p = .80, Chi-squared — A priori threshold of <.05
Statistical Analysis 3: Comparison: Contingency Management vs Placebo; Analysis for 12 month follow-up; Test type: Superiority; p = .12, Chi-squared — A priori threshold of <.05

ADVERSE EVENTS:
Groups:
- Baseline: Placebo: Participants complete urine and breath screens 2 times per week for 8 weeks with no reinforcement for negative results.
Arm/Group | Contingency Management | Baseline
Serious Adverse Events (participants affected / at risk) | 49/165 | 53/165
Other Adverse Events (participants affected / at risk) | 0/165 | 0/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Contingency Management (N=165) | Baseline (N=165)
Death (General disorders) | 4 | 1
Hospitalization (General disorders) | 24 (45) | 26 (39)
Hospitalization (Psychiatric disorders) | 27 (41) | 30 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes